CLINICAL TRIAL: NCT03593798
Title: Lifestyle Intervention and Physical Capacity in Patients With Morbid Obesity
Acronym: LEICO
Status: Completed | Type: Observational
Sponsor: Sykehuset i Vestfold HF (Other)
Collaborators: University college of south-east Norway (Unknown)
Responsible Party: Principal Investigator, Jarle Berge, Principal investigator, Sykehuset i Vestfold HF
Other Study IDs: LEICO
Record Dates: First submitted 2018-04-30; First posted 2018-07-20 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Physical Capacity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Lifestyle — Lifestyle intervention an effect on weight and physical capacity

SUMMARY:
Lifestyle intervention and physical capacity in patients with morbid Obesity (LEICO)

DETAILED DESCRIPTION:
It is still uncertainty about which is the most effective lifestyle treatment to reducing body weight and increased quality of life. Increased physical capacity and muscle mass lead to increased energy expenditure, thus explaining parts of the difference in weight loss achieved after lifestyle treatment. However, literature in this area is limited and need better documentation of how, and to what extent increased physical capacity can affect the effect of lifestyle treatment offered to patients in the health service.

ELIGIBILITY:
Inclusion Criteria:

* Treatment morbidly obese patients (BMI ≥ 40 kg/m2 or BMI 35 to 39.9 kg/m2 with ≥ 1 co morbidity) attending the Vestfold Hospital Trust.

Exclusion Criteria:

* Uncompensated heart failure
* Recent myocardial infarction or stroke (<½ years)
* Severe arrhythmia or heart failure
* Unstable angina pectoris
* Renal failure
* Severe eating disorders
* Active substance abuse

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Obese patient seeking lifestyle intervention program
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2013-11-01 (Actual); Primary Completion 2016-05-30 (Actual); Study Completion 2016-05-30 (Actual)

PRIMARY OUTCOMES:
Weight change at 1-year follow up | Changes from baseline body weight at 1-year follow up.
  Can physical capacity before start of a routine medical care have a impact on weight loss at 1-year follow-up.
  Body weight was measured with patients wearing light clothing and no shoes on Scanvaegt DS-530 (Århus, Denmark) at baseline and after 1-year follow up.
  Changes from baseline body weight at 1-year follow up.
  Participants receive interventions as part of routine medical care, and studie the effect of the intervention.
Weight change at 12-weeks follow up | Changes from baseline body weight at 12-weeks follow up.
  Can physical capacity before start of a routine medical care have a impact on weight loss at 12-weeks follow-up.
  Body weight was measured with patients wearing light clothing and no shoes on Scanvaegt DS-530 (Århus, Denmark) at baseline and after 12-weeks follow up.
  Changes from baseline body weight at 12-weeks follow up.
  Participants receive interventions as part of routine medical care, and studie the effect of the intervention.

SECONDARY OUTCOMES:
Physical capacity changes after 12 weeks as assessed by the maximal oxygen uptake test | Changes from baseline physical capacity at 12-weeks follow up.
  Can the mean twelve-week change in physical capacity be associated with weight loss.
  The maximal oxygen uptake test was performed as an incremental treadmill test on Woodway ELG 55 (Waukesha, Germany) or, for patients with walking restrictions, on an incremental bicycle test (Lode Corival V3, Lode BV, Groningen, Netherlands). Oxygen uptake was registered using the Jaeger oxycon pro ergospirometry test system (Jaeger Oxycon Pro JLAB 5.x, Hoechberg, Germany).
  Changes from baseline physical capacity at 12-weeks follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Hertel, PhD, Study Director — The Hospital of Vestfold
Locations (2):
- Norway (2):
  - Telemark University College, Bø
  - Vestfold Hospital Trust, Tønsberg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Berge J, Storen O, Hertel JK, Gjevestad E, Smastuen MC, Hjelmesaeth J. Associations between cardiorespiratory fitness and weight loss in patients with severe obesity undergoing an intensive lifestyle intervention program: retrospective cohort study. BMC Endocr Disord. 2019 Jul 1;19(1):69. doi: 10.1186/s12902-019-0394-z. PMID 31262301

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-05): https://cdn.clinicaltrials.gov/large-docs/98/NCT03593798/Prot_SAP_000.pdf